CLINICAL TRIAL: NCT00647660
Title: Single-Dose Fasting Bioequivalence Study of Nadolol/Bendroflumethiazide Tablets (80 mg/5 mg; Mylan) to Corzide® Tablets (80 mg/5 mg; King) in Healthy Volunteers
Brief Title: Fasting Study of Nadolol/Bendroflumethiazide Tablets 80 mg/5 mg and Corzide® Tablets 80 mg/5 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullivan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NABE-0626
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Nadolol; Bendroflumethiazide

ARMS (2):
- 1 (Experimental): Nadolol/Bendroflumethiazide Tablets 80 mg/5 mg
  Interventions: Drug: Nadolol/Bendroflumethiazide Tablets 80 mg/5 mg
- 2 (Active Comparator): Corzide® Tablets 80 mg/5 mg
  Interventions: Drug: Corzide® Tablets 80 mg/5 mg

INTERVENTIONS:
Drug: Nadolol/Bendroflumethiazide Tablets 80 mg/5 mg — 80/5mg, single dose fasting
  Arms: 1
Drug: Corzide® Tablets 80 mg/5 mg — 80/5mg, single dose fasting
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's nadolol/bendroflumethiazide 80 mg/5 mg tablets to King's Corzide® 80 mg/5 mg tablets following a single, oral 80 mg/5 mg (1 x 80 mg/5 mg) dose administered under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older
2. Sex: Male and/or non-pregnant, non-lactating female

   1. Women of childbearing potential must have negative serum beta human chorionic gonadotropin (β-HCG) pregnancy tests performed within 21 days prior to the start of the study and on the evening prior to each dose administration. If dosing is scheduled on weekends, serum for the HCG pregnancy test can be collected within 48 hours prior to dosing for each study period. An additional serum (β-HCG) pregnancy test will be performed upon completion of the study.
   2. Women of childbearing potential must practice abstinence or use an acceptable form of contraception throughout the duration of the study. Acceptable forms of contraception include the following:

      1. hormonal contraceptives taken throughout the study, or
      2. intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
      3. barrier methods containing or used in conjunction with a spermicidal agent, or
      4. surgical sterility (tubal ligation, oophorectomy or hysterectomy) or postmenopausal accompanied with a documented postmenopausal course of at least one year.
   3. Hormonal replacement therapy will be allowed in this study
   4. Women will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

      1. postmenopausal with an absence of menses for at least one (1) year, or
      2. bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
      3. total hysterectomy
   5. During the course of the study, from study screen until study exit, all men and women of childbearing potential must use a spermicide-containing barrier method of contraception in addition to their current contraceptive device. This requirement should be documented in the informed consent form.
3. Weight: At least 60 kg (132 lbs.) for men and 48 kg (106 lbs.) for women and all subjects having a Body Mass Index (BMI) greater than or equal to 19 but less than or equal to 30 (see Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
4. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, 12-lead ECG, hepatitis B and hepatitis C tests, HIV test, and urine drug screen including amphetamine, benzodiazepine, cannabinoid, cocaine, opiate screen, phencyclidine, and methadone) performed within 21 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco products within 1 year of the start of the study.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. Positive test for any drug included in the urine drug screen.
   6. History of drug and/or alcohol abuse.
3. Medications:

   1. Use of any prescription or over-the-counter (OTC) medications within the 14 days prior to the initial dose of study medication (other than hormonal contraceptives and hormone replacement therapy)
   2. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, or neurologic disease.
   2. Acute illness at the time of either the pre-study medical evaluation or dosing.
   3. A positive HIV, hepatitis B, or hepatitis C test result.
   4. A history of asthma, bronchospastic disease, chronic bronchitis, sinus bradycardia, and greater than 1st degree conduction block.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
6. Bradycardia less than 50 beats/minute in the supine position, as measured by ECG, at the screening visit or prior to Period I Day 1 dosing.
7. Sitting pulse rate of less than 60 beats per minute and a sitting systolic blood pressure less than 90 or greater than 140 or a sitting diastolic blood pressure less than 60 or greater than 90 after a five-minute resting period at the Screening Visit or prior to Period I Day 1 dosing.
8. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
9. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
10. Allergy or hypersensitivity to nadolol, propranolol, or other β-adrenergic receptor blockers, bendroflumethiazide, sulfonamide-derived drugs, thiazides, or other related products.
11. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
12. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D., Principal Investigator — PRACS Institute Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html